CLINICAL TRIAL: NCT03521128
Title: A Randomized Trial Comparing Radiological Tubal Blockage Versus Laparoscopic Salpingectomy in Infertile Women With Hydrosalpinx During in Vitro Fertilization Treatment
Brief Title: Comparing Radiological Tubal Blockage Versus Laparoscopic Salpingectomy in Infertile Women With Hydrosalpinx During in Vitro Fertilization Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment, no participants enrolled
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-04
Record Dates: First submitted 2018-04-12; First posted 2018-05-11 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: IVF-ET; Hydrosalpinx

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the radiological tubal blockage group (Experimental)
  Interventions: Procedure: radiological tubal blockage
- the laparoscopic salpingectomy group (Active Comparator)
  Interventions: Procedure: laparoscopic salpingectomy

INTERVENTIONS:
Procedure: radiological tubal blockage — In radiological tubal blockage group, under the fluoroscopy of X-ray, after confirming HX by HSG, selective catheterization will be done for the affected tube and micro spring coils will be put in to the interstitial tube and isthmus through micro catheter. The micro spring coil will be placed into the proximal end of the Fallopian tube (unilateral or bilateral depending on whether one or two HX were present) through micro catheter under the fluoroscopy of X-ray. Then HSG will be carried out to check the position of the micro spring coil and confirm complete blockage. Four weeks after the radiological procedure, a HSG will be performed to recheck the position of the micro spring coil and complete blockage of the tubes. FET is proceeded in the next menstrual cycle after HSG examination.
  Arms: the radiological tubal blockage group
Procedure: laparoscopic salpingectomy — In the laparoscopic salpingectomy group, after confirming HX, a unilateral or bilateral salpingectomy will be performed in a standard manner, depending on whether unilateral or bilateral HX are present. In women with extensive pelvic adhesions during laparoscopy, proximal tubal ligation will be performed as an alternative procedure to salpingectomy. FET is proceeded in the next menstrual cycle after the laparoscopic operation.
  Arms: the laparoscopic salpingectomy group

SUMMARY:
Hydrosalpinx (HX) has a detrimental effect on the rates of implantation, pregnancy, live delivery, and early pregnancy loss during in vitro fertilization (IVF). The effectiveness of radiological tubal blockage has not been compared with the standard treatment of laparoscopic salpingectomy in randomized trials. The investigators aim in this randomized trial to compare the live birth rate of radiological tubal blockage versus laparoscopic salpingectomy in infertility women with HX prior to frozen-thawed embryo transfer (FET). Eligible women will be recruited and randomized into one of the following two groups: (1) the radiological tubal blockage group and (2) the laparoscopic salpingectomy group. The primary outcome is the live birth rate.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-43 years at the time of IVF/ICSI treatment
* Unilateral or bilateral HX visible on pelvic ultrasound or hysterosalpingogram
* At least one frozen embryo or blastocyst available for transfer

Exclusion Criteria:

* A history of pelvic inflammatory disease within 6 months
* HX that were already blocked proximally on hysterosalpingogram
* Frozen pelvis from previous laparoscopy
* Women with fibroids interfering with radiological tubal blockage
* Undergoing preimplantation genetic testing

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
live birth rate | a live birth after 22 weeks gestation, through study completion, an average of 1 year
  the rate of live births per cycle

SECONDARY OUTCOMES:
positive hCG level | A blood hCG test is performed 14 days after the FET, up to 14 days
  defined with the result of serum β-hCG ≥10 mIU/mL.
clinical pregnancy rate | presence of intrauterine gestational sac on ultrasound at 6 weeks of pregnancy, up to 6 weeks
  presence of intrauterine gestational sac on ultrasound at 6 weeks of pregnancy
ongoing pregnancy rate | iable pregnancy beyond gestation 12 weeks, up to 12 weeks
  presence of a fetal pole with pulsation at 12 weeks of gestation
implantation rate | number of gestational sacs per embryo transferred at 6 weeks of pregnancy, up to 6 weeks
  number of gestational sacs per embryo transferred
multiple pregnancy | multiple pregnancy beyond gestation 12 weeks up to 12 weeks
  more than one intrauterine sacs on scanning
miscarriage rate | a clinically recognized pregnancy loss before the 22 weeks of pregnancy, up to 22 weeks
  defined as a clinically recognized pregnancy loss before the 22 weeks of pregnancy. The denominator is the clinical pregnancy.
ectopic pregnancy | ectopic pregnancy during first trimester, up to 12 weeks
  pregnancy outside the uterine cavity
birth weight | a live birth after 22 weeks gestation, through study completion, an average of 1 year
  birth weight of the baby delivered

CONTACTS AND LOCATIONS:
Locations (1):
- ShangHai JIAI Genetics&IVF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared. Data will be available when beginning 3 months and ending 5 years following article publication. To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with.Data will be made available by the following way. Proposals should be directed to lihe198900@163.com. And data are available for 5 years at a third party website (link to be included after the article publication).
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Aboulghar MA, Mansour RT, Serour GI. Controversies in the modern management of hydrosalpinx. Hum Reprod Update. 1998 Nov-Dec;4(6):882-90. doi: 10.1093/humupd/4.6.882. PMID 10098478
- [Background] Camus E, Poncelet C, Goffinet F, Wainer B, Merlet F, Nisand I, Philippe HJ. Pregnancy rates after in-vitro fertilization in cases of tubal infertility with and without hydrosalpinx: a meta-analysis of published comparative studies. Hum Reprod. 1999 May;14(5):1243-9. doi: 10.1093/humrep/14.5.1243. PMID 10325271
- [Background] Li Q, Kuang YP, Yang HL, Fu YL, Sun H, Fan LP, Shi HB. [Application of fallopian tube embolization before in vitro fertilization and embryo transfer dealing with the hydrosalpinx]. Zhonghua Fu Chan Ke Za Zhi. 2008 Jun;43(6):414-7. Chinese. PMID 19035133
- [Background] Xu B, Zhang Q, Zhao J, Wang Y, Xu D, Li Y. Pregnancy outcome of in vitro fertilization after Essure and laparoscopic management of hydrosalpinx: a systematic review and meta-analysis. Fertil Steril. 2017 Jul;108(1):84-95.e5. doi: 10.1016/j.fertnstert.2017.05.005. Epub 2017 Jun 1. PMID 28579408
- [Background] Arora P, Arora RS, Cahill D. Essure((R)) for management of hydrosalpinx prior to in vitro fertilisation-a systematic review and pooled analysis. BJOG. 2014 Apr;121(5):527-36. doi: 10.1111/1471-0528.12533. Epub 2014 Jan 3. PMID 24393165
- [Background] Johnson N, van Voorst S, Sowter MC, Strandell A, Mol BW. Surgical treatment for tubal disease in women due to undergo in vitro fertilisation. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD002125. doi: 10.1002/14651858.CD002125.pub3. PMID 20091531